CLINICAL TRIAL: NCT07245914
Title: A Consumer Health Study Evaluating the Impact of Pivit on Weight Loss and Appetite in Overweight Individuals
Status: Active, not recruiting | Type: Observational
Sponsor: Olfactive Biosolutions, Inc. (Industry)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS16
Record Dates: First submitted 2025-09-15; First posted 2025-11-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Obesity &Amp;Amp;Amp; Overweight; Obesity (Body Mass Index &Amp;Amp;Amp;Amp;gt;30 kg/m2)
Keywords: obesity; overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Product Group: All 125 study participants will be receiving the study product, Pivit, throughout the course of the study. There is no placebo group for this study.
  Interventions: Dietary Supplement: The Study Product (Pivit)

INTERVENTIONS:
Dietary Supplement: The Study Product (Pivit) — All 125 study participants will be taking the study product, Pivit, throughout the course of the study. There is no placebo intervention for this study.

SUMMARY:
The purpose of this study is to observe the impact of Pivit on body weight in overweight individuals. Additionally, the study aims to observe the impact of the product on appetite, hunger, cravings, and general well-being via activities and technologies that can successfully and effectively be completed in a home setting. A consumer-driven, decentralized observational clinical research study is therefore well-suited for examining the impact of this product in this population.

The study team will examine the outcomes in a broad age-range of adults who have chosen to try this product. The study will incorporate participant reported outcome questionnaires and surveys and at-home body weight measurement using a personal scale. There is no "doctor-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the product and take part in the observational process with self-reported measures and at-home body weight measurement. Findings from this study will contribute knowledge toward the tolerability and formulation of the plant-derived consumer product and the design of future studies.

DETAILED DESCRIPTION:
Pivit is a proprietary and patented formulation of food molecules, designed to act on receptors in the gut to cause a natural secretion of GLP-1 and GIP hormones. GLP-1 and GIP are hormones that naturally delay stomach emptying to reduce appetite and trigger the pancreas to secrete insulin which regulates blood sugar. Pivit has been shown to naturally increase GLP-1 and GIP in human cellular studies and in initial consumer trials, which in turn increase feelings of satiety and lessen hunger pangs, lower blood sugar and support healthy insulin sensitivity. Pivit may also lessen interest in alcohol and reduce 'food noise,' thoughts about food throughout the day and curtail the urge to snack.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Has self-reported body mass index (BMI) between 25 and 34.9 kg/m2.
* Interested in learning about weight management and appetite and in trying Pivit product for themselves.
* GLP-1 medication naive or has not taken any GLP-1 inducing weight-loss medications prior to enrollment.
* Willingness to refrain from taking any weight loss supplements during the study.
* Has a personal digital weight scale at home to use during the study.
* In good general health at the time of screening (Investigator discretion).
* Able to read and understand English.
* Able to read, understand, and provide informed consent.
* Able to use a personal smartphone device and download Chloe by People Science.
* Able to receive shipment of the product at an address within the United States.
* Able to complete study assessments over the course of up to 17 weeks.

Exclusion Criteria:

Any potential participants who:

* Do not have a personal smartphone, internet access, or unwilling to download Chloe.
* Currently on or planning to start a fad diet, keto diet, pure carnivore diet, raw food diet, fruitarian diet, liquid diet (does not include vegans or vegetarians)

Concomitant Conditions and Therapies:

* Any investigational therapies or treatments within 30 days prior to enrollment.
* GLP-1 receptor agonists and related incretin mimetics, (e.g. semaglutide (Ozempic, Rybelsus), dulaglutide (Trulicity), exenatide (Byetta, Bydureon), liraglutide (Victoza, Saxenda), lixisenatide (Adlyxin), sitagliptin (Januvia, Janumet), saxagliptin (Onglyza, Komblglyze), alogliptin (Nesina, Kazano, Oseni), linagliptin (Tradjenta, Jentadueto) or tirzepatide (Mounjaro)
* Currently diagnosed with Alcohol Use Disorder and/or Substance Use Disorder
* Currently pregnant, planning to become pregnant in the next 1 month, or breastfeeding
* Any underlying medical conditions or comorbidities that may confound the evaluation of the study outcomes.
* Have a significant illness, disease or condition which, in the opinion of the principal investigator, may impact their ability to participate in the study or impact the study outcomes.
* Known hypersensitivity or previous allergic reaction to Cinnamaldehyde, Spearmint Oil, Eugenol, Butyl butyryl lactate, Benzyl acetate, Lauric acid, Sodium-Copper Chlorophyllin, Sunflower Seed Oil, Gelatin, Glycerin
* Are unlikely for any reason to be able to comply with the trial or considered unsuited for participation in the study by the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants must be 18 years or older, have a body mass index between 25 and 34.9, glucagon-like peptide-1 (GLP1) naive, and interested in trying Pivit, the study product, for themselves.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 weeks; 3 months
  The primary outcome measure for this study will be to observe the impact of the study product, Pivit, on individual weight. This will be measured by assessing the change from baseline in body weight after three months of study product use.

SECONDARY OUTCOMES:
BMI | 12 weeks ; 3 months
  Another outcome measure for this study will be to observe the impact of the study product, Pivit, on body mass index (using reported weight and height). This will be measured by assessing the change from baseline in body mass index after three months of study product use.
Gastrointestinal Symptoms | 12 weeks; 3 months
  A secondary outcome measure will be to assess the impact of the study product, Pivit, on gastrointestinal symptoms. This will be measured by assessing the change from baseline in Gastrointestinal Symptom Questionnaire score after 12 weeks of product use (Likert scale: Absent - I did not have this symptom at all Mild - I had this symptom occasionally, but it did not really bother me Moderate - I had this symptom often, it bothered me quite a bit Severe - I had this symptom very often, it bothered me a great deal), with a lower value indicating a better outcome.
Gastrointestinal Symptoms | 12 weeks; 3 months
  A secondary outcome measure will be to assess the impact of the study product, Pivit, on gastrointestinal symptoms. This will be measured by assessing the change from baseline in average scores on gastrointestinal symptoms including stomach discomfort, constipation, bloating, diarrhea, food noise, lightheadedness, and sweating after 12 weeks of product use using a 10-point VAS with 0 being absent and 10 being severe.
Cognition and Behavior | 12 weeks; 3 months
  The secondary outcome will be to assess the impact of Pivit on cognitive and behavioral components of eating. This will be assessed using the change from baseline using the Three Factor Eating Questionnaire (TFEQ) score after 12 weeks of product use. The TFEQ is a 4 point scale (Definitely true, Mostly true, Mostly false, Definitely false) with a lower score indicating a better outcome.
General Health and Well-Being | 12 weeks; 3 months
  A secondary outcome will be to assess the impact of the study product, Pivit, on individual appetite, hunger, cravings, night-time snacking and general well-being. This will be measured by a 5 point visual analog scale with 0 - strongly disagree to 5 - strongly agree, assessing the change from baseline in average weekly questionnaire scores for appetite, hunger and general after three months of product use.
Adverse Events | 12 weeks ; 3 months
  The final secondary outcome will be to observe the safety and tolerability of the study product, Pivit. This will be measured by an assessment of the number, frequency, and severity of adverse events (AEs), serious adverse events (SAEs) and adverse event withdrawals reported over the study period of 12 weeks / 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, MD, Principal Investigator — People Science, Inc.
Locations (1):
- People Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
This will need to be discussed internally.